CLINICAL TRIAL: NCT04276532
Title: Sentinel Lymph Node Sampling Versus Systematic Pelvic Lymphadenectomy on the Prognosis for Patients With Middle-high Risk Endometrial Cancer Confined to the Uterus Before Surgery: a Non-inferiority Randomized Controlled Trial
Brief Title: Sentinel Lymph Node Sampling for Patients With Middle-high Risk Endometrial Cancer Confined to the Uterus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Collaborators: Fudan University (Other); Tongji Hospital (Other); West China Second University Hospital (Other); Sun Yat-sen University (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Vice President of Obstetrics and Gynecology Hospital of Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01 2019-12
Record Dates: First submitted 2020-02-13; First posted 2020-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Middle-high Risk Endometrial Cancer; Sentinel Lymph Node Sampling; Prognosis
Keywords: Middle-high risk endometrial cancer; Sentinel lymph node sampling; Pelvic lymphadenectomy; Prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sentinel lymph node sampling (Experimental): Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus sentinel lymph node sampling (SLN)
  Interventions: Procedure: sentinel lymph node sampling (SLN)
- Pelvic lymphadenectomy (Active Comparator): Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus pelvic lymphonodectomy (PLN) with para-aortic sampling
  Interventions: Procedure: pelvic lymphonodectomy (PLN)

INTERVENTIONS:
Procedure: sentinel lymph node sampling (SLN) — Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus sentinel lymph node sampling (SLN).
  1. The principles of surgery procedures and post-operative adjuvant therapies will follow the latest NCCN guidelines；
  2. Surgery carried out by laparotomy, laparoscope, or robotic surgery are accepted；
  3. Colored dyes including indocyanine green (ICG) (preferred), methylene blue, carbon nanotube for sentinel lymph node are accepted.
  Arms: Sentinel lymph node sampling
Procedure: pelvic lymphonodectomy (PLN) — Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus pelvic lymphonodectomy (PLN) with para-aortic sampling
  Arms: Pelvic lymphadenectomy

SUMMARY:
Aim To investigate the effect of sentinel lymph node (SLN) sampling on the prognosis of patients with middle-high risk endometrial cancer obviously confined to the uterus before surgery.

DETAILED DESCRIPTION:
Aim to investigate the effect of sentinel lymph node (SLN) sampling on the prognosis of patients with middle-high risk endometrial cancer obviously confined to the uterus before surgery.

Rationale The diagnostic value of sentinel lymph node sampling has been widely approved. NCCN guideline suggested that "SLN mapping can be considered for the surgical staging of apparent uterine-confined malignancy when there is no metastasis demonstrated by imaging studies or no obvious extrauterine disease at exploration". However, the role of SLN in the prognosis of mid-high risk endometrial cancer clinically confined to the uterus is unclear. There are big concerns that SLN sampling only without lymph node dissection might miss isolated para-aortic lymph node metastasis or remain lymph node with metastasis other than SLN unremoved and thus affect the prognosis of patients. NCCN also suggested that "Para-aortic nodal evaluation from the inframesenteric and infraenal regions may also be utilized for staging in women with high-risk tumors such as deeply invasive lesions, high-grade histology, and tumors of serous carcinoma, clear cell carcinoma or carcinosarcoma. Thus, it is necessary to carry out a randomized trail to investigate the role of SLN in the prognosis of middle-high risk endometrial cancer obviously confined to the uterus before surgery.

Ethnics This study were approved by the Ethics Committees of Obstetrics and Gynecology Hospital of Fudan University and all other institutes. Before initiation of study procedures, written informed consent will be obtained from each patient regarding risks of treatments and agreement of using their clinical data for research purpose.

Randomization and Treatment This is a multicentered, open-label, randomized clinical trial. Randomization will be carried out in each center. A computer-based procedure of simple randomization (SPSS for Mac, version 22.0; IBM ) will be used for participant enrollment and randomization. Before an individual is successfully enrolled, her treatment assignment will remain concealed. This trial will be open label: patients and study physicians were aware of treatment assignment.

Eligible patients in each center will be randomly assigned (1:1) to receive:

1. Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus pelvic lymphonodectomy (PLN) with para-aortic sampling, or 2. Total hysterectomy with/without bilateral salpingooophorectomy (THBO) plus sentinel lymph node sampling (SLN).

1. The principles of surgery procedures and post-operative adjuvant therapies will follow the latest NCCN guidelines.
2. Surgery carried out by laparotomy, laparoscope, or robotic surgery are accepted.
3. Colored dyes including indocyanine green (ICG) (preferred), methylene blue, carbon nanotube for sentinel lymph node are accepted.
4. Postoperative adjuvant treatments are carried out following the latest NCCN guidelines according to doctors' choice.

Statistical analyses On the basis of data from previous studies (GOG249, FRACOGYN), the 2-year PFS is expected to be 88% in the PLN group and 87% in SLN group. SLN would be considered as inferior to PLN if the 2-year PFS in SLN group is higher than 80%. An accrual of 780 patients in 3 years will provide the study with adequate power (80%) to detect a clinically relevant absolute difference of 8% in 2-year PFS (88% vs 80%) between both groups (one-sided test, a=0.025), with a lost follow up rate ≤10% . Analyses will be done firstly by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old;
2. Clinically diagnosed (by pre-surgical pathology and radiology) as primary endometrial cancer confined to uterus with middle-high risk factors:

   1. Disease limited to the uterus on image study (MRI, CT or ultrasound);
   2. including all histological types of endometrial cancer (endometrioid, serous, clear cell, carcinosarcoma, and undifferentiated carcinoma); not including uterine sarcoma
   3. excluding low-risk endometrial cancer (endometrioid G 1-2 with pre-surgical endometrial lesion≤2cm and myometrial invasion <50%);
   4. with one or more middle-high risk factors including: endometrioid endometrial cancer G3, myometrial invasion ≥50%, tumor size≥2cm, type II endometrial cancer; LVSI
   5. diagnosis should be confirmed by at least two senior clinicians.
3. Be able to undergo staging surgery.

Exclusion Criteria:

1. During pregnancy or perinatal period;
2. With malignancies other than endometrial cancer;
3. With history of important organs transplantation;
4. With immune diseases requiring taking immunosuppressants
5. With severe mental illness or brain function disorders
6. With history of drug abuse;
7. Allergic to contrast agent;
8. Still participating in other clinical trials;
9. Not willing to accept surgery or trial protocol;
10. Not eligible for surgery;
11. Had hysterectomy, chemotherapy, radiotherapy, or hormone therapy before the trail;
12. Had retroperitoneum lymph node dissection for other reasons.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 780 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2030-02-12 (Estimated)

PRIMARY OUTCOMES:
The 2-year progression-free survival (2-year PFS) | 2 years
  The percentage of patients who have first relapse within 2 years after surgery (SLN or LND)

SECONDARY OUTCOMES:
The 5-year PFS | 5 years
  The percentage of patients who have first relapse within 5 years after surgery (SLN or LND)
The 5-year overall survival (OS) | 5 years
  The percentage of patients who die within 5 years after surgery (SLN or LND)
Adverse effect and quality of life (QOL) | Adverse effect: during the surgery, 30 days after surgery; QQL: 1 month before surgery, 6 months, 12 months after surgery
  The occurence rate of each adverse effects related to surgery (SLN or LND, the scores of each QOL survay

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Guan J, Xue Y, Zang RY, Liu JH, Zhu JQ, Zheng Y, Wang B, Wang HY, Chen XJ. Sentinel lymph Node mapping versus systematic pelvic lymphadenectomy on the prognosis for patients with intermediate-high-risk Endometrial Cancer confined to the uterus before surgery: trial protocol for a non-inferiority randomized controlled trial (SNEC trial). J Gynecol Oncol. 2021 Jul;32(4):e60. doi: 10.3802/jgo.2021.32.e60. PMID 34085796